CLINICAL TRIAL: NCT01549535
Title: Polyp Detection With The Peerscope System™: A Randomized Tandem Colonoscopy Study
Brief Title: Polyp Detection With The Peerscope System™
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PeerMedical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: CD-1158
Record Dates: First submitted 2012-02-13; First posted 2012-03-09 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Colon Polyps and Adenomas; Colon Cancer
MeSH Terms: conditions — Colonic Polyps; Adenoma; Colonic Neoplasms | interventions — Colonoscopy; Mass Screening

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Group A (study group) (Active Comparator): Subjects in Group A (study group) will undergo a Standard view colonoscopy followed immediately by a PeerScope System™ extended view colonoscopy.
  Interventions: Device: Colonoscopy done with:PeerMedical System and Olympus/Pentax/Fuji colonoscopy system
- Group B (control group) (Active Comparator): Group B (control group) will undergo a PeerScope System™ extended view colonoscopy followed immediately by a Standard view colonoscopy.
  Interventions: Device: Colonoscopy done with:PeerMedical System and Olympus/Pentax/Fuji colonoscopy system

INTERVENTIONS:
Device: Colonoscopy done with:PeerMedical System and Olympus/Pentax/Fuji colonoscopy system — endoscopic diagnosis, treatment and video observation of the digestive tract, endoscopy and endoscopic treatment within the lower digestive tract (including the anus, rectum, sigmoid colon, colon and ileocecal valve) of adults patients
  Other Names: Colonoscopy; Polyp detection; Screening

SUMMARY:
The PeerScope System consists of Peer Medical camera heads, endoscopes, video system, light source and other ancillary equipment. The system is intended for endoscopic diagnosis, treatment and video observation of the digestive tract. The PeerScope system model B is indicated for use for endoscopy and endoscopic treatment within the lower digestive tract (including the anus, rectum, sigmoid colon, colon and ileocecal valve) of adults patients.

Objective:To compare the additional diagnostic yield obtained by using the PeerScope System™ extended view vs. the diagnostic yield obtained by the Standard view colonoscopy.

In addition, time measurements including time to cecum, time for withdrawal and overall procedure time will be analyzed and reported for each group.

DETAILED DESCRIPTION:
Design:

Patients who are scheduled for screening, surveillance or diagnostic colonoscopy will be recruited to the study and randomized to one of two groups. Each enrolled subject will undergo two "back-to-back" procedures.

Subjects in Group A (study group) will undergo a Standard view colonoscopy followed immediately by a PeerScope System™ extended view colonoscopy. Subjects in Group B (control group) will undergo a PeerScope System™ extended view colonoscopy followed immediately by a Standard view colonoscopy.

Results from the two groups will be analyzed and compared, with primary outcome measures being detection rates for total polyps and detection rates for adenomas. Secondary outcome measures will include withdrawal time, total procedure time and characteristics of polyps detected, including size and histological results.

Subjects will be followed through a 24 hour and a 7 days telephone interview for analysis of unexpected adverse events. Clinical results will be analyzed using various statistical measures of significance.

Study Design:

Multi-center study with up to 196 patients. No. of Patients:

Up to 196 treated patients will be enrolled into the study. Primary Performance Endpoint:

* Standard view colonoscopy adenoma overall detection rate compared to the extended view overall adenoma detection rate using the PeerScope System™
* Standard view colonoscopy overall polyp detection rate compared to the extended view overall polyp detection rate using the PeerScope System™.

Safety Analysis:

Incidence of device-related and procedure-related serious adverse events. Incidence of complications using PeerScope System™

Known complications include:

* Perforation;
* Severe abdominal pain;
* Infection;
* Bleeding (other than expected minor bleeding due to therapeutic procedures e.g. polypectomy);
* Inducing inflammation of diverticulum
* Arrhythmia, bradycardia, hypotension, hypoxia
* Death

Secondary Endpoints / Other Outcomes:

1. Performance of therapeutic interventions, such as biopsies, polypectomies, APC etc.
2. Procedure time. The following will be recorded: a. Time for intubation to the cecum. b. Time for withdrawal from the cecum to the anal verge. c. Total procedure time A stopwatch will be used for stopping the timing of the procedure for any polypectomy performed and then restarting once the polypectomy is completed, meaning that purely procedure time is measured
3. Sedation dosage
4. Patient satisfaction. Patient's pain at the end of the procedure will be recorded using VAS scale. Results of 24 hour telephone follow-up to assess for post-procedural patient satisfactory will be recorded on the CRF.

Inclusion criteria:

* Subject between the ages of 18 and 70
* The patient is undergoing colonoscopy for screening, for surveillance in follow-up of previous polypectomy or for diagnostic workup;
* Written informed consent must be available before enrollment in the trial
* For women with childbearing potential, adequate contraception

Exclusion criteria:

* Patients with a history of colonic resection;
* Patients with known (or newly diagnosed) inflammatory bowel disease;
* Patients with a personal history of polyposis syndrome;
* Patients with suspected chronic stricture potentially precluding complete colonoscopy;
* Patients with diverticulitis or toxic megacolon;
* Patients with a history of radiation therapy to abdomen or pelvis;
* Patients with acute lower GI bleeding
* Patients who are currently enrolled in another clinical investigation in which the intervention might compromise the safety of the patient's participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subject between the ages of 18 and 70
* The patient is undergoing colonoscopy for screening, for surveillance in follow-up of previous polypectomy or for diagnostic workup;
* Written informed consent must be available before enrollment in the trial
* For women with childbearing potential, adequate contraception

Exclusion Criteria:

* Patients with a history of colonic resection;
* Patients with known (or newly diagnosed) inflammatory bowel disease;
* Patients with a personal history of polyposis syndrome;
* Patients with suspected chronic stricture potentially precluding complete colonoscopy;
* Patients with diverticulitis or toxic megacolon;
* Patients with a history of radiation therapy to abdomen or pelvis;
* Patients with acute lower GI bleeding
* Patients who are currently enrolled in another clinical investigation in which the intervention might compromise the safety of the patient's participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2012-02; Primary Completion 2013-03 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
polyp detection rate | 1 year
  Sample size calculation is based on detecting a difference in the adenoma overall detection rate and the overall polyp detection rate using the PeerScope System™ extended view as compared to Standard view colonoscopy.
  Total sample size will be 196 patients. Each patient will undergo the procedure by the two devices: PeerScope System™ extended view and Standard view colonoscopy. The rational for this sample size is based on detecting a rate difference of 20% between the study devices.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Gralnek, Prof., Principal Investigator — Rambam Health Care Campus; Peter Siersema, Prof., Principal Investigator — UMC Utrecht; Erwin Santo, Prof., Principal Investigator — The Tel Aviv Sourasky Medical Center; Ori Segol, Dr., Principal Investigator — Carmel Medical Center; Alan Sloyer, Dr., Principal Investigator — North Shore Gastroenterology Associates, P.C.; Jay S. Fenster, Dr., Principal Investigator — Southshore Gasstroenterology, P.C
Locations (6):
- United States (2):
  - North Shore Gasstroenterology Assoiates, P.C., New York, New York
  - Southshore Gasstroenterology, P.C, New York, New York
- Israel (3):
  - Carmel Medical Center, Haifa
  - Elisha Medical Center, Haifa
  - The Tel Aviv Sourasky Medical Center, Tel Aviv
- UMC, Utrecht, Netherlands

REFERENCES:
- [Derived] Gralnek IM, Siersema PD, Halpern Z, Segol O, Melhem A, Suissa A, Santo E, Sloyer A, Fenster J, Moons LM, Dik VK, D'Agostino RB Jr, Rex DK. Standard forward-viewing colonoscopy versus full-spectrum endoscopy: an international, multicentre, randomised, tandem colonoscopy trial. Lancet Oncol. 2014 Mar;15(3):353-60. doi: 10.1016/S1470-2045(14)70020-8. Epub 2014 Feb 20. PMID 24560453